CLINICAL TRIAL: NCT03793439
Title: Tofacitinib Hypothesis-generating, Pilot Study for Corticosteroid-Dependent Sarcoidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jim Rosenbaum, Professor of Ophthalmology, Medicine, and Cell Biology, OHSU, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017902
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Sarcoidosis, Pulmonary; Sarcoidosis Lung; Sarcoidosis
Keywords: Sarcoidosis; Corticosteroid dependent sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — tofacitinib; Tablets; Clinical Trials as Topic; Spirometry; Respiratory Function Tests; Sequence Analysis, RNA; Clinical Laboratory Techniques; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Open-label, interventional, proof of concept, hypothesis-generating study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label treatment (Experimental): All subjects will receive tofacitinib 5mg twice daily from week 0 to week 16, and a corticosteroid taper starting at week 16. Participants also undergo spirometry, RNA sequence testing, and laboratory evaluations.
  Interventions: Drug: Tofacitinib 5mg Oral Tablet [Xeljanz] 16 week trial; Diagnostic Test: Spirometry; Genetic: RNA Sequencing; Diagnostic Test: Laboratory testing; Drug: Corticosteroid; Drug: Tofacitinib 5mg [Xeljanz] 1 year open-label extension

INTERVENTIONS:
Drug: Tofacitinib 5mg Oral Tablet [Xeljanz] 16 week trial — Tofacitinib 5mg oral table twice daily for 16 weeks
  Other Names: Xeljanz; tofacitinib
Diagnostic Test: Spirometry — Spirometry testing at baseline, week 4, week 8, week 12, and week 16
  Other Names: Pulmonary function test
Genetic: RNA Sequencing — RNA sequencing test at baseline and week 16
Diagnostic Test: Laboratory testing — Laboratory testing at baseline and weeks 2, 4, 8, 12 and 16
  Other Names: Blood work
Drug: Corticosteroid — Taper corticosteroids starting at week 4
  Other Names: Corticosteroid taper; Prednisone taper; Steroid taper
Drug: Tofacitinib 5mg [Xeljanz] 1 year open-label extension — After 16 weeks, subjects who meet the primary end-point will be permitted an optional one year open-label extension.
  Other Names: tofacitinib; Xeljanz

SUMMARY:
This is a pilot study to determine whether further research is warranted to assess whether tofacitinib is an effective steroid sparing treatment for pulmonary sarcoidosis. The primary endpoint for this study is a 50% or greater reduction in corticosteroid requirement.

DETAILED DESCRIPTION:
Primary Objectives:

Objective 1: Test the hypothesis that the addition of tofacitinib will allow patients with sarcoidosis to have 50% or greater reduction in their corticosteroid requirement without a significant decrease in pulmonary function testing, and with a similar quality of life as measured by a validated questionnaire (1).

Objective 2: Test the hypothesis that the addition of tofacitinib will result in significantly decreased expression of signal transducer and activator of transcription (STAT)-1 dependent gene expression.

Outline:

This is a 16-week open-label, interventional, proof of concept, hypothesis-generating study. All subjects will receive Tofacitinib 5mg twice daily for 16 weeks. After four weeks on Tofacitinib, the corticosteroid will be tapered per a pre-defined protocol; once a reduction of 50% has been achieved, any further taper will be per physician discretion. After 16 weeks, subjects who meet the primary end-point will be permitted an optional one year open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Meet World Association of Sarcoidosis and other Granulomatous Disorders (WASOG) definition of pulmonary sarcoid
* Histologically proven sarcoid
* Evidence of pulmonary sarcoid on chest radiograph
* Forced vital capacity of > 50%
* Require 15-30mg/day of prednisone or equivalent corticosteroid to control sarcoidosis.
* Stable dose of prednisone or equivalent corticosteroid for 4 weeks prior to enrollment.

Exclusion Criteria:

* May be taking methotrexate but not other immunosuppressive or immunomodulatory treatments in the two months prior to study period. This includes but is not limited to azathioprine, cyclophosphamide, leflunomide, mycophenolate mofetil, cyclosporine, tacrolimus, and biologic medications.
* Patients requiring >30mg/day prednisone or equivalent.
* Pregnant or lactating women.
* Hemoglobin < 9g/dL or hematocrit < 30%
* White blood cell count <3.0 K/cu mm
* Absolute neutrophil count <1.2 K/cu mm
* Platelet count <100 K/cu mm
* Subjects with an estimated glomerular filtration rate (GFR) ≤40 ml/min
* Subjects with a total bilirubin, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal at screening.
* Severe, progressive, or uncontrolled chronic liver disease including fibrosis, cirrhosis, or recent or active hepatitis.
* History of any lymphoproliferative disorder such as Epstein Barr virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggest of current lymphatic disease.
* Current malignancy or history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis and aspergilloma, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Have a known infection with human immunodeficiency virus (HIV)
* Have current signs and symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac (New York Heart Association class III or IV), neurologic, or cerebral diseases (with the exception of sarcoidosis).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Rosenbaum, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 1, 2022 until December 31, 2023
Access Criteria: Email friedmam@ohsu.edu

REFERENCES:
- [Background] Rosenbaum JT, Choi D, Wilson DJ, Grossniklaus HE, Harrington CA, Sibley CH, Dailey RA, Ng JD, Steele EA, Czyz CN, Foster JA, Tse D, Alabiad C, Dubovy S, Parekh P, Harris GJ, Kazim M, Patel P, White V, Dolman P, Korn BS, Kikkawa D, Edward DP, Alkatan H, Al-Hussain H, Yeatts RP, Selva D, Stauffer P, Planck SR. Parallel Gene Expression Changes in Sarcoidosis Involving the Lacrimal Gland, Orbital Tissue, or Blood. JAMA Ophthalmol. 2015 Jul;133(7):770-7. doi: 10.1001/jamaophthalmol.2015.0726. PMID 25880323
- [Derived] Friedman MA, Le B, Stevens J, Desmarais J, Seifer D, Ogle K, Choi D, Harrington CA, Jackson P, Rosenbaum JT. Tofacitinib as a Steroid-Sparing Therapy in Pulmonary Sarcoidosis, an Open-Label Prospective Proof-of-Concept Study. Lung. 2021 Apr;199(2):147-153. doi: 10.1007/s00408-021-00436-8. Epub 2021 Apr 7. PMID 33825964

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: Tofacitinib 5 mg twice daily by mouth
Period: Overall Study
Arm/Group | Open Label
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 5 participants were analyzed for baseline characteristics. The overall number of baseline participants did not differ from the number assigned to arms and entire study.
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 40.8 [35 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% Reduction in Corticosteroid Requirement
Description: 50% reduction in corticosteroid requirement by week 16, without significant decline in their pulmonary function-defined as a >15% decline in forced vital capacity (FVC), forced expiratory volume at 1 second (FEV1), or diffusing capacity of lung for carbon monoxide (DLCO) relative to the baseline value
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Open Label: open label tofacitinib
Arm/Group | Open Label
Number analyzed (Participants) | 5
Participants | 3

2. Secondary Outcome: Number of Participants With Significantly Decreased Expression of STAT1 Mediated Genes as Determined by RNA Sequencing
Description: Peripheral blood RNA sequencing performed before and after 16 weeks of tofacitinib treatment. Significant changes are defined as at least 1.5 fold change in the expression of STAT1-mediated genes, with a false discover rate p value of < 0.05.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from week 0 (start of study drug) until study drug was stopped, plus 4 weeks of post-treatment follow up. This corresponded to 72 weeks for subjects who completed the study and open-label extension: study (16 weeks), open-label extension (52 weeks), and post-treatment follow up (4 weeks). Adverse event data from subjects who terminated the study early were collected until study drug was stopped + 4 weeks.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=5)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) — Flare of neurosarcoidosis with peripheral neuropathy requiring escalation of glucocorticoids and subsequent withdrawal from the clinical trial. Treated with high dose glucocorticoids and infliximab, resolved.
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) — Upper extremity cellulitis during post-study monitoring period. Occurred while on prednisone 30 mg/day, 9 days after the last study drug dose, 10 days after infliximab 5 mg/kg, resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) — Mild rash on scalp and face, resolved without intervention.
Vomiting (Gastrointestinal disorders) | 1 (1) — Emesis after suspected ingestion of spoiled food, resolved without intervention.
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. ER visit, arthrocentesis with non-inflammatory fluid, no crystals, resolved with conservative management. 2. Motor vehicle accident w/ ER visit for right knee and left shoulder pain. X-rays without fracture. Resolved with physical therapy
Diarrhea (Gastrointestinal disorders) | 1 (1) — 3 days of diarrhea, resolved without intervention.
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Exacerbation of seasonal nasal allergies
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough up to 3-4x/week, resolved without intervention.
Renal colic (Renal and urinary disorders) | 1 (1) — ER visit for renal colic, initially thought to be urinary tract infection and given antibiotic however urinalysis and culture negative. Renal stones on CT, required pain medication and hydration, resolved.
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — ER visit for bronchitis, no pneumonia in imaging. Treated with oral antibiotics, resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03793439/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT03793439/ICF_001.pdf